CLINICAL TRIAL: NCT06893666
Title: Effects of Play Based Therapy on Attention Level of Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0678
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Down Syndrome
Keywords: Play Therapy; Down Syndrome; Attention; Randomized Control Trial; Child Development
MeSH Terms: conditions — Down Syndrome | interventions — Play Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Play based therapy (Experimental): Experimental group was given pay based therapy. Total of 4 sessions were given each session of 40min.
  Interventions: Other: Play based therapy
- Child centered play therapy (Active Comparator): Control group was given child centered play therapy. Total of 4 sessions were given each session of 40min.
  Interventions: Other: Child centered play therapy

INTERVENTIONS:
Other: Play based therapy — Experimental group was given pay based therapy. Total of 4 sessions were given each session of 40min.
  Arms: Play based therapy
Other: Child centered play therapy — Control group was given child centered play therapy. Total of 4 sessions were given each session of 40min.
  Arms: Child centered play therapy

SUMMARY:
The aim of the study is to examine the attention level of children with down syndrome receiving play based therapy as compared to children receiving child centered play therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age: 3-5 years
* Gender: Both male and female
* Children who are currently taking speech therapy sessions with parental involvement.
* Medically stable children with no severe ongoing health issues that could interfere with their participation in the study.

Exclusion Criteria:

* Children with severe sensory impairments
* Co-morbid neurological conditions that may confound the results
* Children who received intervention from any other institute

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
NHS Attention and Listening Screener | Baseline and 4 weeks
  The screener was designed to measure attention and listening of children. It is dichotomous (yes/no) comprising of 9 items according to age rang of 3-5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Aleena Irum, Ms-SLP, Principal Investigator — Riphah International University
Locations (1):
- Aleena Irum, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu WP, Tsai WH, Lin LY, Hong RB, Hwang YS. The Beneficial Effects of Massage on Motor Development and Sensory Processing in Young Children with Developmental Delay: A Randomized Control Trial Study. Dev Neurorehabil. 2019 Oct;22(7):487-495. doi: 10.1080/17518423.2018.1537317. Epub 2018 Oct 30. PMID 30376388
- [Background] Manshi, Dimple Choudhry, Anshu Kumari, & Priyanka Gulati. (2023). To Compare the Attention Span of Down Syndrome Children with Healthy Children of Same Age Group. International Journal of Medical Science and Diagnosis Research, 7(2). https://doi.org/10.32553/ijmsdr.v7i2.976